CLINICAL TRIAL: NCT00358761
Title: Investigation of Southern Tick-Associated Rash Illness (STARI)
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060207; 06-I-0207
Record Dates: First submitted 2006-07-29; First posted 2006-08-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-12-11

CONDITIONS: Southern Tick-Associated Rash Illness
Keywords: Lone Star Tick; Borrelia; Skin Biopsy; Spirochete; Erythema Migrans; Southern Tick-Assoicated Rash Illness; STARI
MeSH Terms: conditions — Southern tick-associated rash illness; Lyme Disease; Glossitis, Benign Migratory

SUMMARY:
This study will evaluate blood and tissue samples for a condition called Southern Tick-Associated Rash Illness (STARI). This is a skin rash resembling erythema migrans, the rash found in people infected with Lyme disease. In the south and southeastern United States, STARI is associated with the bite of the lone star tick. Researchers seek a better understanding of the cause of STARI. Through researchers' knowledge, diagnostic tests could be developed. NIH is conducting this study along with the Centers for Disease Control and Prevention (CDC).

Patients ages 14 years and older who have recently been diagnosed with possible STARI, who have not taken antibiotics for it longer than 1 day, and whose skin does not form large scars may be eligible for this study. About 20 participants will be enrolled over a 5-year period. Patients will visit the NIH Clinical Center for two or three visits. The first visit may last 2 hours. Photographs will be taken of the rash, and a blood sample of about 1-1/2 tablespoons will be collected for tests. Patients will undergo a punch biopsy of three small pieces of skin, from the rash. The area of the skin will be cleaned, and patients will receive a local anesthetic at the biopsy site. A sharp instrument will remove a round plug of skin, about the size of half a pencil eraser. Patients may feel a pushing sensation, but there should not be pain. The site usually heals without sutures, though the doctors may close it with special adhesive bandages or one or two sutures. Patients will receive instructions about how to take care of the biopsy site. If sutures are used, patients will return in 7 to 10 days to have them removed-or a patient's own doctor may remove the sutures. Patients will return to NIH at 4 to 6 weeks following their first visit. At that time, they will answer questions about how they are doing and donate about 2 tablespoons of blood. Blood and skin samples will be used for research at NIH and CDC.

...

DETAILED DESCRIPTION:
Southern Tick-Associated Rash Illness (STARI) is a rash similar to the rash of Lyme disease that occurs in persons residing in southeastern and south-central states and is associated with the bite of the lone star tick, Amblyomma americanum. The cause of the rash is unknown, as it is the natural course of the disease. This protocol aims to investigate the cause of STARI, in conjunction with the Center for Disease Control and Prevention (CDC). Skin biopsies and blood samples will be taken from patients with suspected STARI and will be used to search for an infectious agent and to develop diagnostic tests for the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Enrolled in protocol 02-I-0055.

A person who is at least 14 years old.

Acute onset (within 14 days of visit to NIH) of an annular, erythematous, expanding erythema migrans (EM)-like rash that attains a size of at least 5 cm in diameter, when no alternative explanation for the rash can be found, and thought by the study physician to have a high likelihood to be due to STARI (due to exposure history, tick identification).

History of tick bite at the rash site, or potential exposure to ticks in the southeastern and south central United States within 14 days prior to rash onset (including Maryland and Virginia).

Consent to storage of biologic samples for later testing.

EXCLUSION CRITERIA:

A person who, in the judgment of the investigator, would be at increased risk from the skin biopsy procedure and unlikely to be able to mount a serological response to the agent (for example, bone marrow transplant, B cell deficiency).

EXCLUSION FROM SKIN BIOPSY PORTION OF STUDY:

A person who meets the case definition but whose EM-like rash occurs on the face, neck, scalp, or over the tibia will not be enrolled for purposes of obtaining a skin biopsy specimen. Such a person may enroll for purposes of providing a clinical history and blood samples only. This exclusion also applies to patients with a history of forming large thick scars after skin injuries or surgery, or who have a history of excessive bleeding after cuts or procedures or are taking anticoagulants, or have severe skin disease. Also, patients who have received more than 24 hours of antibiotic treatment for the rash will be excluded from the biopsy. Patient with a history of allergy to lidocaine will also be excluded from the biopsy portion of the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-07-20; Study Completion 2012-12-11

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Varela AS, Luttrell MP, Howerth EW, Moore VA, Davidson WR, Stallknecht DE, Little SE. First culture isolation of Borrelia lonestari, putative agent of southern tick-associated rash illness. J Clin Microbiol. 2004 Mar;42(3):1163-9. doi: 10.1128/JCM.42.3.1163-1169.2004. PMID 15004069
- [Background] James AM, Liveris D, Wormser GP, Schwartz I, Montecalvo MA, Johnson BJ. Borrelia lonestari infection after a bite by an Amblyomma americanum tick. J Infect Dis. 2001 Jun 15;183(12):1810-4. doi: 10.1086/320721. Epub 2001 May 17. PMID 11372036
- [Background] Campbell GL, Paul WS, Schriefer ME, Craven RB, Robbins KE, Dennis DT. Epidemiologic and diagnostic studies of patients with suspected early Lyme disease, Missouri, 1990-1993. J Infect Dis. 1995 Aug;172(2):470-80. doi: 10.1093/infdis/172.2.470. PMID 7622891